CLINICAL TRIAL: NCT06704347
Title: A Phase 1, Open-Label Study Assessing the Safety, Pharmacokinetics, Pharmacodynamics, and Biomarkers of Single Ascending Dose Regimens of XT-150 for the Treatment of Amyotrophic Lateral Sclerosis (ALS)
Brief Title: Safety Study of XT-150 in Participants With ALS
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Xalud Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XT-150-1-0402
Record Dates: First submitted 2024-11-20; First posted 2024-11-26 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: 1.5 mg XT-150 (Experimental): Participants will be administered 1.5 mg of XT-150 once by intrathecal injection on Day 1. An intrathecal injection is an injection using a thin needle inserted into the spinal canal at the base of your spinal cord performed by your study doctor.
  Interventions: Biological: XT-150
- Cohort 2: 4.5 mg XT-150 (Experimental): Participants will be administered 1.5 mg of XT-150 once by intrathecal injection on Day 1. An intrathecal injection is an injection using a thin needle inserted into the spinal canal at the base of your spinal cord performed by your study doctor.
  Interventions: Biological: XT-150

INTERVENTIONS:
Biological: XT-150 — XT-150 is a small piece of plasmid DNA (genetic material) that produces a variant of the anti-inflammatory cytokine, Interleukin 10 (IL-10).

SUMMARY:
This is a Phase 1, open-label, multi-center safety study of XT-150 in adult participants with Amyotrophic Lateral Sclerosis (ALS).

Participants providing informed consent and meeting all study eligibility criteria will be enrolled in the study and will receive a single injection of XT-150 at the Baseline visit. Follow-up visits will occur over 180 days (6 months) after the injection.

8 participants (4 participants per dose level) will be enrolled sequentially in up to 2 ascending, single dose cohorts: Cohort 1: 1.5 mg XT-150 Cohort 2: 4.5 mg XT-150

DETAILED DESCRIPTION:
The main questions this study is aiming to answer are:

* What adverse events are reported during this study? An adverse event is any "side effect" that participants have during a study. Adverse events may or may not be caused by XT-150. The study doctors will check participants' ALS and general health throughout the trial.
* Does XT-150 have any effects on participants' physical examination findings, vital signs, or laboratory values?

In addition to evaluating the safety of XT-150, this study will also collect samples to provide information on the following:

* The levels of XT-150 in your body
* The effect of XT-150 on cytokines including interleukin (IL)-10
* The effect of XT-150 on relevant ALS biomarkers such as Neurofilament Light (NfL)

In addition, ALS functional score, breathing capacity and strength will be collected over the course of the study.

ELIGIBILITY:
Key Inclusion Criteria:

* Adults between 18 and 80 years of age
* Male or female, if of childbearing potential or sexually active, strict contraception required
* Have ALS diagnosed by a doctor (specifically, sporadic or familial ALS diagnosed as clinically probable, lab-supported probable or definite ALS defined by the El Escorial criteria)
* Have had symptoms of ALS (muscle weakness) within 36 months of starting this study
* Have the ability to slowly exhale a volume of air at least 60% of what is expected for the participant's sex, height and age
* Have not received treatment for ALS or are currently on a stable dose of an approved treatment for ALS. Patients currently receiving Tofersen are not eligible.
* Able to receive the study injection intrathecally, determined by the study doctor
* Able to undergo the study procedures and adhere to the study visit schedule at the time of study entry, with an estimated life expectancy of 6 months or greater

Key Exclusion Criteria:

* Have an implanted shunt to drain cerebrospinal fluid (CSF) or an implanted CNS catheter
* Have an implanted of diaphragm pacing system
* Tracheostomy
* History or current diagnosis of cardiac conditions or ECG abnormalities indicating significant risk of safety for participants in the study
* History or current diagnosis of respiratory conditions such as COPD
* History or current diagnosis of cancer, chemical meningitis, HIV, Hep B, Hep C, uncontrolled diabetes
* Presence of an autoimmune condition (for example, rheumatoid arthritis or lupus) requiring treatment or immunodeficiency
* Clinical or laboratory evidence of hepatic or renal disease/injury.
* Taking any prohibited medications
* Women who are pregnant or nursing
* Use of any investigational drugs or devices within 30 days or 5 half-lives of the study agent (whichever is longer). Exception: Observational, non-interventional clinical studies are allowed in the opinion of the study doctor.
* Any other condition that the study doctor feels could compromise the participant's safety, ability to communicate with the study staff, or the quality of the data

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants reporting adverse events (AEs), Serious Adverse Events (SAEs) and AEs of Special Interest (AESIs) | Up to Day 180
Number of participants with clinically significant physical examination findings | Up to Day 180
Number of participants with clinically significant vital sign abnormalities | Up to Day 180
  Vital signs include temperature, heart rate, respiratory rate and blood pressure
Number of participants with clinically significant laboratory abnormalities | Up to Day 180
  Clinical laboratory assessments include hematology, chemistry, coagulation, lipids, C-reactive protein, erythrocyte sedimentation rate and CSF total protein, cell count and glucose

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Barrow Neurological Institute (St. Joseph's), Phoenix, Arizona
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford Health, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: No